CLINICAL TRIAL: NCT04716530
Title: The Changing Panorama in Risk Factors of Cerebral Palsy: A Single National Tertiary Center Experience
Brief Title: The Changing Panorama in Risk Factors of Cerebral Palsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Bilinç Doğruöz Karatekin, Principal Investigator, Istanbul Medeniyet University
Other Study IDs: Istanbul MU CP
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; etiology; risk factors; low birth weight; prematurity
MeSH Terms: conditions — Cerebral Palsy; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- born before 2000: No patient treatment is associated with the study.
  Interventions: Other: No intervention is associated with the study.
- born between 2000-2010: No patient treatment is associated with the study.
  Interventions: Other: No intervention is associated with the study.
- born after 2010: No patient treatment is associated with the study.
  Interventions: Other: No intervention is associated with the study.

INTERVENTIONS:
Other: No intervention is associated with the study. — No intervention is associated with the study.

SUMMARY:
The study will be carried of scanning the database of 296 individuals with cerebral palsy followed in the university pediatric rehabilitation clinic. Cerebral palsy risk factors and demographic information will be obtained from the database. The data will be classified according to date of birth, divided into 3 groups: those born before 2000, those born between 2000-2010, and those born after 2010.Changes in cerebral palsy risk factors will be investigated at 10-year intervals.

DETAILED DESCRIPTION:
The study will be carried of scanning the database of 296 individuals with cerebral palsy followed in the university pediatric rehabilitation clinic. Cerebral palsy risk factors and demographic information will be obtained from the database.

Cerebral palsy subtypes classified according to The Surveillance for Cerebral Palsy in Europe (SCPE) classification into four groups: spastic (unilateral and bilateral), dyskinetic (dystonic and choreoathetoic), ataxic/hypotonic, non-classifiable. Cerebral palsy risk factors will be primarily divided into 4 as preconceptional, antenatal, intrapartum and neonatal risk factors. Then, risk factors in the data will be distributed to the appropriate risk factor group.

The data will be classified according to date of birth, divided into 3 groups: those born before 2000, those born between 2000-2010, and those born after 2010. Changes in cerebral palsy risk factors will be investigated at 10-year intervals.

ELIGIBILITY:
Inclusion Criteria:

* cerebral palsy patients

Exclusion Criteria:

* missing data on the cerebral palsy database

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in our cerebral palsy database
Sampling Method: Non-Probability Sample
Enrollment: 296 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-02-20 (Estimated)

PRIMARY OUTCOMES:
Define the risk factors of cerebral palsy | 1 month
  Risk factors of cerebral palsy questioned as preconceptional, antenatal, intrapartum and neonatal.
Define the change in the risk factors among age groups | 1 month
  The difference in cerebral palsy risk factors in age groups measured by chi-square statistics (born before 2000/ born between 2000-2010/ born after 2010)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University Faculty of Medicine, Physical Medicine and Rehabilitation Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No